CLINICAL TRIAL: NCT05844319
Title: THE EFFECT OF PAIN MANAGEMENT TRAINING ON ACTIVITIES OF DAILY LIVING AND QUALITY OF LIFE IN KNEE OSTEOARTHRITIS
Brief Title: Pain Management In Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTANBULC4
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Osteoarthritis; Knee Osteoarthritis; Pain, Chronic
Keywords: Osteoarthritis; Pain Management; Activities of Daily Living; Quality of Life; Tele-education
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): Following the completion of the evaluations of the cases, the following 6-step program will be applied to cope with the pain:
  1. Informative education about the disease
  2. Teaching relaxation positions for pain management
  3. Relaxation exercises with breathing exercises
  4. Training on ergonomic approaches in daily life (correct sitting, lying, working, carrying, etc.)
  5. Education of principles of joint protection
  6. Creating and training a personalized physical activity and exercise plan
  Interventions: Other: tele-education

INTERVENTIONS:
Other: tele-education — The treatment of the patients will be carried out by tele-education method.

SUMMARY:
In this study, it was aimed to investigate the effect of pain management education in individuals with knee osteoarthritis with chronic pain.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA), also known as degenerative joint disease of the knee, is typically the result of wear and tear and progressive loss of joint cartilage. Knee osteoarthritis can be divided into two types, primary and secondary. It is most common in the elderly. The intensity of clinical symptoms can vary from person to person. However, they typically become more severe, more frequent, and more debilitating over time. The rate of progression also varies with each individual. People suffering from knee osteoarthritis complain of limited range of motion and pain when they move their knee or start walking. In advanced disease, they may complain of nocturnal or persistent knee pain and the functionality of the joint is severely impaired. Knee osteoarthritis treatment begins with non-surgical (conservative) treatment methods. Non-surgical treatment includes patient education, lifestyle modification, and the use of orthotic devices. It has been shown that untreated pain in the elderly can have a general impact on their quality of life and lead to depression, anxiety, social isolation, cognitive impairment, inactivity, and sleep disorders. The aim of our project is to provide training for patients diagnosed with knee osteoarthritis with chronic pain to be able to control their pain with self-management and to perform activities of daily living more easily. Appropriate knowledge and awareness can improve their quality of life. Performing safe and accurate pain management practices in the elderly can improve their performance, quality of life, increase their comfort and reduce their care costs. In this study, it was aimed to investigate the effect of pain management education in individuals with knee osteoarthritis with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with knee OA according to the criteria of the American College of Rheumatology (ACR)
* Be between 45 and 75 years old
* Stage 2-3 according to Kellgren Lawrence (K-L) in the radiological examination

Exclusion Criteria:

* Having active synovitis
* Receiving physical therapy in the last 6 months
* People with neurological problems that affect walking
* Those with arthritis in the ankle and hip joint
* Those with serious respiratory, central, peripheral, vascular and uncontrolled metabolic problems that will prevent exercise.
* Have had surgery on the lower extremity in the past
* Intra-articular steroid injections in the last 6 months
* Use of psychoactive drugs

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | on the first day and eighth week change
  We will use the Knee Injury and Osteoarthritis Outcome Score (KOOS) in order not to exceed the pain and daily life span of our patients. It is a scale that evaluates the functional status and groups related to knee injuries and knee osteoarthritis. Other definition of pain has 5 subgroups, including functional status related to daily life span, functional status in sports and leisure activities, and sequence-related quality of life. It consists of 42 questions lasting approximately 10 minutes. Each subscale is scored between 0-100. 0 indicates serious problem, 100 indicates no problem. A score of 10 and above indicates that it changes clinically.

SECONDARY OUTCOMES:
The McGill Pain Questionnaire | on the first day and eighth week change
  We will use the McGill Pain Questionnaire to evaluate the pain status of our patients. The McGill Pain Questionnaire is a chart with descriptive words about pain. Words are normally divided into four main categories: sensory, emotional, evaluative, and miscellaneous. Within these categories are specific subcategories that contain words used to describe the intensity of a particular sensation or emotional response. Following a particular method, patients choose the most appropriate words from each category to describe their pain to their doctor as precisely and precisely as possible. This can lead to better pain management and, in some cases, better and faster diagnosis. The most common version has 20 subcategories of descriptive words.
Short Form-12 | on the first day and eighth week change
  Similar to SF-36, SF-12 has physical functionality (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functionality (1 item) It consists of 8 sub-dimensions and 12 items: emotional role (2 items) and mental health (2 items). Items related to physical and emotional role were answered as dichotomy (yes or no), while other items had Likert type options ranging between 3 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET YAZGAN, BSc, Study Director — Istanbul University - Cerrahpasa; MELIKE KARAVUL, BSc, Principal Investigator — Istanbul University - Cerrahpasa; HUSEYIN BAYBAS, BSc, Principal Investigator — Istanbul University - Cerrahpasa; ELA TARAKCI, Prof, Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Tugba Civi Karaaslan, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No